CLINICAL TRIAL: NCT00502125
Title: A Pilot Study: In Vivo Reflectance Confocal Imaging for Detection of Neoplasia of Oral Mucosa
Brief Title: In Vivo Confocal Imaging of Oral Mucosa
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: ID02-494
Record Dates: First submitted 2007-07-13; First posted 2007-07-17 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Oral Tumors
Keywords: Reflectance Confocal Imaging; Oral Mucosal Lesions; Oral Mucosa Disease; Neoplasia Detection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue samples will be removed.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with oral lesions
  Interventions: Procedure: Reflectance Confocal Imaging

INTERVENTIONS:
Procedure: Reflectance Confocal Imaging — A photograph will be taken of any abnormal areas inside the mouth. A small probe will expose the oral lining to a small amount of light. Some of this light will be reflected back into the probe, and be picked up by a computer. Pictures will be made of the tissue.

SUMMARY:
The objective of this study is to evaluate the feasibility of using reflectance confocal imaging to noninvasively detect and diagnose oral dysplasia and early carcinoma.

DETAILED DESCRIPTION:
The study will take place at M. D. Anderson. Examinations will be performed in the cancer prevention, head and neck or dental clinics, or the operating room for patients who get scheduled for surgery as part of their standard care.

Abnormal looking areas (lesions) inside the mouth may be a sign of cancer or changes that may lead to cancer. Researchers are looking for a practical way to tell early on whether these lesions are cancer or may become cancer. This study will look at a technique called reflectance confocal imaging.

Participants in this study will have an examination of the mouth. A photograph will be taken of any abnormal areas inside the mouth. Then a small probe, about the size of a large ink pen, will be placed gently against one to two abnormal appearing areas, and one normal appearing area inside the mouth. The probe will expose the oral lining to a small amount of light. Some of this light will be reflected back into the probe, and be picked up by a computer. Pictures will be made of the tissue.

A small amount of vinegar will be placed at each site with a cotton swab before the probe is placed. The procedure takes about 1-2 minutes at each site. A small sample of tissue from each site, both the normal and abnormal, will be removed. The biopsies done on the normal tissue are done for this study only and are not part of standard care. The samples will be removed either at the time of surgery or under local anesthesia in the clinic. Briefly, the small areas to be biopsied will be numbed with topical anesthesia and an injection of local anesthesia. Then a small amount of tissue, about as big as a pencil eraser, will be removed with sterile surgical instruments. This should cause little discomfort or bleeding. The tissue will be placed in a special fluid and then looked at with a special microscope. The tissue samples will be examined with a microscope by a pathologist to learn if the tissue is cancerous or precancerous. These results will be compared with the pictures that were made of the lining of the mouth.

You will not be told of any of the experimental findings. The pathology review of the tissue removed will be available to the treating physician for patient care.

THIS IS AN INVESTIGATIONAL STUDY. The device used for reflectance confocal imaging is an investigational device. It is considered a non-significant risk device by the FDA to be used for research only. A total of 22 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* Patients with oral lesions who give informed consent to participate in the study.
* Any person with an oral lesion, particularly those suspicious for dysplasia or carcinoma.

Exclusion Criteria:

* Lack of any oral mucosal lesions
* Oral lesions not physically accessible for probe placement or biopsy
* Unwillingness to tolerate probe placement, dilute acetic acid rinse or biopsy
* Unwillingness to provide informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with oral lesions.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2003-01; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
To study if using reflectance confocal imaging can detect and diagnose abnormal growths in the mouth and early cancer. | 6 Years

CONTACTS AND LOCATIONS:
Overall Officials: Ann M. Gillenwater, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org